CLINICAL TRIAL: NCT00397553
Title: Multicenter, Open, Non-randomised Phase III Clinical Study of Efficacy and Safety of Insulin Glulisine Injected Subcutaneously in Patients With Type 1 Diabetes Mellitus Using Also Insulin Glargine
Brief Title: Insulin Glulisine, Diabetes Mellitus Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3517
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine

ARMS (1):
- Insulin Glulisine (Experimental)
  Interventions: Drug: Insulin glulisine

INTERVENTIONS:
Drug: Insulin glulisine

SUMMARY:
To provide local data on efficacy and safety of insulin glulisine in patients with Type 1 Diabetes Mellitus receiving insulin glargine as basic insulin therapy

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, Type 1
* HbA1c 6.5-11.0%
* BMI <35 kg/m²

Exclusion Criteria:

* Diabetes mellitus, Type 2

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 52 weeks

SECONDARY OUTCOMES:
HbA1c | 26 weeks
Fasting Blood Glucose | 26 weeks
Fasting Blood Glucose | 52 weeks
Post-prandial glycemia (2 hour after breakfast) | 26 weeks
Post-prandial glycemia (2 hour after breakfast) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marina Atarshchikova, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Moscow, Russia